CLINICAL TRIAL: NCT05138809
Title: Evaluation of the Lakeshore Online Fitness Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Lakeshore Foundation (Other)
Responsible Party: Principal Investigator, Tapan Shirish Mehta, Associate Professor and Director of Research, Department of Health Services Administration, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300007405; 90REGE000 (Other Grant/Funding Number: NIDILRR)
Record Dates: First submitted 2021-09-02; First posted 2021-12-01 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Physically Disabled
Keywords: Exercise; Physical Activity; Virtual Exercise; Mobility Impairment
MeSH Terms: conditions — Motor Activity | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Exercise (Experimental): Use online exercise platform
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — Use online exercise platform

SUMMARY:
The purpose of this project is to test feasibility of an online platform that delivers virtual exercise programs for individuals with physical disabilities.

DETAILED DESCRIPTION:
The sample pool of this study is members of a community fitness center that serves individuals with physical disabilities and chronic health conditions. The study will be advertised to the members through flyers, newsletters, social media, and center's website.

Members logging into the center's online exercise system will be presented with a brief introduction to the study and asked if they would like to "Opt In" to receive further information. When the system receives on Opt In trigger, the member will be asked a series of eligibility screening questions regarding their age, fluency in English, and whether or not they have a mobility limitation or problems with gait, balance, and/or coordination. Members who are not eligible will be directed back to center's online exercise system for regular access to the program options. Members who are eligible will be asked to complete an e-Consent form. Members who decline consent will be directed back to the center's online exercise system for regular access to the program options. Members who accept consent will be provided with a welcome page listing next steps.

After review of the welcome page, participants will be asked to complete a series of online surveys that will be completed before and after 8 weeks of participation. All surveys, except for the health history, are composed of Likert-scale questions. After the participant completes all the surveys, the system will trigger a message to the research staff to schedule an onboarding call with the participant to provide an overview of the system and available online classes (live and pre-recorded). Participants will be encouraged to accumulate a total of 150 minutes of moderate or 75 minutes of vigorous exercise throughout the week.

Participants will then be on their own to participate in virtual classes as they wish. Each time the participant completes a live online class, they will be asked to complete a brief survey to provide their perceptions regarding the class. Compensation in the form of a gift card will be provided to participants for completion of the Pre and Post intervention surveys. In addition, small incentives will be provided to the participants meeting certain participation criteria.

At the end of each week, the research staff will monitor logins and post-class survey responses. In the event that a participant has not logged into the system during the past 7 days or indicates issues via the post class survey a member of the research team will call them. Coaching calls will be made at the end of Week 2, 4, and 6 as needed. If the issue is lack of interest or difficulty with the existing classes, a new series of pre-recorded exercise videos will be made available to the participant for remainder of the eight weeks. This option will only be available once. At the end of the 8 weeks, participants will be asked to complete the survey package again.

ELIGIBILITY:
Inclusion Criteria:

* Must be a member of Lakeshore Foundation
* Age 18 years or above
* Mobility limitation, problem with gait, balance and/or coordination
* Fluency in English

Exclusion Criteria:

* No access to internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2021-09-22 (Actual); Primary Completion 2022-05-02 (Actual); Study Completion 2022-05-02 (Actual)

PRIMARY OUTCOMES:
Change in Level of Physical activity from baseline at 8 weeks | Before and after 8 weeks of participation
  Assess current level of physical activity. Godin Leisure-Time Exercise Questionnaire. Four questions, score ranges from 0 to 119. A higher score indicates higher level of physical activity.

SECONDARY OUTCOMES:
Change in Reasons for exercise from baseline at 8 weeks | Before and after 8 weeks of participation
  Participant's reasons for exercise (survey). Ten questions, response from 1 to 5 for each question (1 = not important, 5 = very important).
Change in Self-efficacy for exercise from baseline at 8 weeks | Before and after 8 weeks of participation
  Participant's belief in their ability to exercise. Self-Efficacy for Exercise Scale. Nine questions. score ranges from 0 to 90. A higher score indicates higher self-efficacy for exercise.
Change in Outcome expectations for exercise from baseline at 8 weeks | Before and after 8 weeks of participation
  What outcomes does the participant expect as a result of exercising. Multidimensional Outcome Expectations for Exercise Scale. Fifteen questions, score ranges from 15 to 75. A higher score indicates higher expectations for exercise outcomes. Also, three subscales: Physical (6 items), Self-evaluation (5 items), and Social (4 items)
Change in Exercise goals/plans from baseline at 8 weeks | Before and after 8 weeks of participation
  Participant's exercise goals and plans. Exercise Goal-Setting and Planning/Scheduling Scales. Ten questions related to goal setting, score ranges from 10 to 50. A higher score indicates higher goal setting. Ten questions related to exercise planning, score ranges from 10 to 50. A higher score indicates greater exercise planning.
Change in Health-related quality of life from baseline at 8 weeks | Before and after 8 weeks of participation
  Participant's self-reported quality of life. Enabled version of the short-form 36 (SF-36E). Thirty-six questions, 8 subscales, two summary scores. The scales are standardized with a scoring algorithm to obtain a score ranging from 0 to 100. Higher scores indicate greater health-related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tapan Mehta, PhD, Principal Investigator — University of Alabama at Birmingham; Mohanraj Thirumalai, PhD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- Lakeshore Foundation, Homewood, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Malone LA, Mehta T, Mendonca CJ, Mohanraj S, Thirumalai M. A prospective non-randomized feasibility study of an online membership-based fitness program for promoting physical activity in people with mobility impairments. Pilot Feasibility Stud. 2024 Aug 2;10(1):104. doi: 10.1186/s40814-024-01528-x. PMID 39095876